CLINICAL TRIAL: NCT03681847
Title: Crystalloids Versus Colloids Versus Hypertonic Saline Co-load During Spinal Anesthesia: Which is More Effective
Brief Title: Crystalloids Versus Colloids Versus Hypertonic Saline as a Co-load During Spinal Anesthesia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ehab Hanafy Shaker, lecturer of anesthesia ,critical care and pain medicine, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ehab-Walaa.Hypertonic
Record Dates: First submitted 2018-09-19; First posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Spinal Anaesthesia
Keywords: hypertonic saline; colloids; normal saline
MeSH Terms: interventions — Saline Solution; Hydroxyethyl Starch Derivatives; Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normal saline (Active Comparator): Patients will receive normal saline 0.9% 15 ml/kg over 15-20 minutes.
  Interventions: Procedure: Normal saline
- Hydroxyethyl starch (Active Comparator): Patients will receive hydroxyethyl starch 130/0.4 in 0.9 % sodium chloride 5 ml/kg over 15-20 minutes.
  Interventions: Procedure: hydroxyethyl starch
- Hypertonic saline (Active Comparator): Patients will receive hypertonic saline 3% (7ml/kg) over 15-20 minutes.
  Interventions: Procedure: Hypertonic saline

INTERVENTIONS:
Procedure: Normal saline — normal saline 0.9% 15 ml/kg over 15-20 minutes.
  Arms: normal saline
Procedure: hydroxyethyl starch — hydroxyethyl starch 130/0.4 in 0.9 % sodium chloride 5 ml/kg over 15-20 minutes.
  Arms: Hydroxyethyl starch
Procedure: Hypertonic saline — hypertonic saline 3% (7ml/kg) over 15-20 minutes.
  Arms: Hypertonic saline

SUMMARY:
Spinal anesthesia is commonly accompanied by hypotension due to vasodilation that follows sympathetic blockade and decreased systemic vascular resistance. Prevention of hypotension is usually achieved through administration of fluids and vasopressors .There is an ongoing debate concerning both the proper fluid timing, pre-load against co-load and fluid type crystalloids against colloids .This study aims at comparing the effectiveness of co-loading of crystalloids versus colloids versus hypertonic saline 3% in preventing hypotension induced by spinal anesthesia.

DETAILED DESCRIPTION:
Spinal anesthesia is commonly accompanied by hypotension due to vasodilation that follows sympathetic blockade and decreased systemic vascular resistance. Prevention of hypotension is usually achieved through administration of fluids and vasopressors . Fluids are either administrated before initiation of spinal anesthesia which is defined as fluid pre-loading or at time of initiation of spinal anesthesia which is defined as fluid co-loading .There is an ongoing debate concerning both the proper fluid timing, pre-load against co-load and fluid type crystalloids against colloids. Fluid preloading with colloids appears to have superior effect on that of crystalloids as the later shows a shorter intravascular half-life. While both colloid and crystalloid co-loading show comparable results .Although crystalloid preloading has been the traditional regimen for long time, it failed to reduce the incidence of hypotension. This is because crystalloids rapidly distribute out of the intravascular compartment to the interstitial space. Superiority of fluid co-loading might be explained by decrease of the extravascular crystalloid redistribution secondary to the simultaneous vasodilatation response to sympathetic block.This study aims at comparing the effectiveness of co-loading of crystalloids versus colloids versus hypertonic saline 3% in preventing hypotension induced by spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* ASA II-III
* Elective lower abdominal surgeries

Exclusion Criteria:

* Coagulation defects
* Abnormal kidney or liver functions
* Local infection at site of injection
* Uncontrolled hypertension
* Bone metastases
* Cardiac disease
* Elevated serum sodium level > 145 mEq/L

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Hypotension | 3 hours
  The development of hypotension

SECONDARY OUTCOMES:
serum sodium level | 3 hours
  measurement of serum sodium level

CONTACTS AND LOCATIONS:
Overall Officials: Ehab H Shaker, MD, Principal Investigator — National Cancer Institute- Cairo University
Locations (1):
- Department of Anesthesia and Pain medicine.National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
after finishing and publishing the study we plan to share it.

REFERENCES:
- See also: Colloid versus Crystallid Co-load with Spinal Anesthesia during Emergent Cesarean Section and Their Effect on Hemodynamic Changes.Lotfy ME; Moustafa AM; Elham M.E, et al. J Am Sci 2014;10(11):158-163] — https://www.ncbi.nlm.nih.gov/pubmed/2528143